CLINICAL TRIAL: NCT04235010
Title: Effects of Genius Toothbrushes on Periodontal Status of Patients Undergoing Fixed Orthodontic Treatment
Brief Title: Genius Toothbrushes on Periodontal Status of Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Serpil Cokakoglu, Assistant Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018DISF007
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Periodontal Inflammation; Toothbrushing; Orthodontic Treatment
Keywords: Genius toothbrush; Orthodontic treatment; Periodontal health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The examiner who performed clinical periodontal parameters was blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual toothbrush (Experimental): Patients used manual orthodontic toothbrush (Oral B Ortho, Procter & Gamble, USA) for four months
  Interventions: Device: Manual toothbrush
- Genius toothbrush (Experimental): Patients used genius orthodontic toothbrush (Oral B Genius 8900, Procter & Gamble, USA) for four months
  Interventions: Device: Genius toothbrush

INTERVENTIONS:
Device: Genius toothbrush — Patients brushed their teeth twice a day for 2 minutes. An integral timer was used in the genius toothbrush group.
  Arms: Genius toothbrush
Device: Manual toothbrush — Patients brushed their teeth twice a day for 2 minutes. During brushing, patients in manual group assigned to use their brushes were provided with a digital timer.
  Arms: Manual toothbrush

SUMMARY:
This study evaluates the effects of genius toothbrushes on periodontal status of patients during fixed orthodontic treatment.Half of the patients received manual orthodontic toothbrushes (Oral B Ortho, Procter & Gamble, USA) with V-shaped bristles and rounded ends. The others received genius orthodontic toothbrush (Oral B Genius 8900, Procter & Gamble, USA) with Oral-B CrossAction brush head, Procter & Gamble, USA).

DETAILED DESCRIPTION:
Powered (genius) toothbrush with position detection technology provides patient to clean all areas of the mouth during the required time. By connecting phone to the Oral-B App, the genius toothbrush uses facial recognition technology to guide patient's brushing, zone to zone. Pressure control and personalization are another characteristics of these toothbrushes. Pressure sensor alerts patient if the brushing is too hard and helps her/him not to put too much pressure by reducing the speed of brush head. Due to the Bluetooth technology, toothbrushing can be performed more efficiently among orthodontic adolescent patients. In addition, the position detection and timer can be used to control which area is brushed in the mouth and how much total brushing time is continued. The application allows patient to see all the days brushing activity and real-time feedback on brushing habits can be received by this way.

ELIGIBILITY:
Inclusion Criteria:

* Permanent dentition with no missing teeth
* No systemic or severe periodontal problems
* Indication of non-extraction fixed orthodontic treatment
* No use of drugs in the past two months
* Absence of physical problems that prevent brushing
* Right handedness for brushing
* Same bracket type (0.022 slot metal, conventional) and ligation technique (wire ligature)
* Finishing of leveling phase (use of rectangular wires)
* Initial total score was between 3 and 10 for the labial surface of each tooth according to the modified Silness and Löe plaque index

Exclusion Criteria:

* Missing teeth
* Systemic or severe periodontal problem
* Indication of extraction treatment
* Use of drugs in the past two months
* Levelling phase of fixed orthodontic treatment

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Löe and Silness gingival index measurement | 1 month
  A score from 0 to 3 is given. Grade 0 indicates normal gingiva; grade 1 mild inflammation with no bleeding; grade 2 moderate inflammation, erythema, swelling, bleeding on probing or when pressure applied; grade 3 severe inflammation, severe erythema and swelling, tendency toward spontaneous hemorrhage, some ulceration
Löe and Silness gingival index measurement | 2 months
  A score from 0 to 3 is given. Grade 0 indicates normal gingiva; grade 1 mild inflammation with no bleeding; grade 2 moderate inflammation, erythema, swelling, bleeding on probing or when pressure applied; grade 3 severe inflammation, severe erythema and swelling, tendency toward spontaneous hemorrhage, some ulceration
Löe and Silness gingival index measurement | 4 months
  A score from 0 to 3 is given. Grade 0 indicates normal gingiva; grade 1 mild inflammation with no bleeding; grade 2 moderate inflammation, erythema, swelling, bleeding on probing or when pressure applied; grade 3 severe inflammation, severe erythema and swelling, tendency toward spontaneous hemorrhage, some ulceration
Modified Silness and Löe plaque index measurement | 1 month
  The buccal surface of each tooth is divided into four zones (mesial, distal, gingival and incisal) to the bracket. Each of the four sites of the buccal tooth surface is given a score from 0 to 3, where 0 indicates the absence of plaque; 1 indicates no plaque visible, but an accumulation of soft deposit on a probe when used to clean the surface; 2 indicates a moderate accumulation of soft deposit on the tooth which can be seen with the naked eye; and 3 indicates an abundance of soft matter on the tooth. For the analysis, values are summed to obtain a total score per participant.
Modified Silness and Löe plaque index measurement | 2 months
  The buccal surface of each tooth is divided into four zones (mesial, distal, gingival and incisal) to the bracket. Each of the four sites of the buccal tooth surface is given a score from 0 to 3, where 0 indicates the absence of plaque; 1 indicates no plaque visible, but an accumulation of soft deposit on a probe when used to clean the surface; 2 indicates a moderate accumulation of soft deposit on the tooth which can be seen with the naked eye; and 3 indicates an abundance of soft matter on the tooth. For the analysis, values are summed to obtain a total score per participant.
Modified Silness and Löe plaque index measurement | 4 months
  The buccal surface of each tooth is divided into four zones (mesial, distal, gingival and incisal) to the bracket. Each of the four sites of the buccal tooth surface is given a score from 0 to 3, where 0 indicates the absence of plaque; 1 indicates no plaque visible, but an accumulation of soft deposit on a probe when used to clean the surface; 2 indicates a moderate accumulation of soft deposit on the tooth which can be seen with the naked eye; and 3 indicates an abundance of soft matter on the tooth. For the analysis, values are summed to obtain a total score per participant.
Bleeding on probing scores | 1 month
  A periodontal probe runs along the marginal gingiva at an angle of approximately 60° to the longitudinal axis of the tooth to determine whether probing elicited marginal bleeding (score 1) or not (score 0). The inflammation was recorded as bleeding scores if bleeding occurred within 30 seconds of probing. Bleeding on probing was estimated as a percentage.
Bleeding on probing scores | 2 months
  A periodontal probe runs along the marginal gingiva at an angle of approximately 60° to the longitudinal axis of the tooth to determine whether probing elicited marginal bleeding (score 1) or not (score 0). The inflammation was recorded as bleeding scores if bleeding occurred within 30 seconds of probing. Bleeding on probing was estimated as a percentage.
Bleeding on probing scores | 4 months
  A periodontal probe runs along the marginal gingiva at an angle of approximately 60° to the longitudinal axis of the tooth to determine whether probing elicited marginal bleeding (score 1) or not (score 0). The inflammation was recorded as bleeding scores if bleeding occurred within 30 seconds of probing. Bleeding on probing was estimated as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University Faculty of Dentistry Department of Orthodontics, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No